CLINICAL TRIAL: NCT05957965
Title: The Effect of Wii Fit Rehabilitation in Patients With Chronic Ankle Instability a Randomized Control Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya abd el hady abbas, principle investigator aya abd el hady abbas, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: clinical trial
Record Dates: First submitted 2023-07-08; First posted 2023-07-24 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Instability, Joint
Keywords: Wii fit rehabilitation; chronic ankle instability; biodex balance system
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise training group (Active Comparator): 30 patients will receive conventional physical therapy training only which consist of strengthening, proprioceptive exercises.
  Interventions: Other: Strengthening, proprioceptive exercises.
- Wii Fit rehabilitation training group (Experimental): 30 patients Wii Fit group will receive Wii Fit rehabilitation training and the same conventional exercise training (strengthening, proprioceptive exercises)
  Interventions: Device: Wii fit; Other: Strengthening, proprioceptive exercises.

INTERVENTIONS:
Device: Wii fit — Nintendo Wii console (Nintendo Co., Ltd, Kyoto, Japan) is the main power unit of Nintendo Wii Fit. Its software includes an interactive video games that is played with a handheld, wireless remote that senses motion and requires the participant to mimic the action of their on - screen character. These games are played using a special Wii balance board in order to perform activities like yoga, balance and aerobics. The Wii remote is the primary controller for Nintendo's Wii console. The motion sensing capability is the main feature of it. It allows the user to interact with and manipulate items on screen via pointing.
  Other Names: Nintendo Wii Fit system
  Arms: Wii Fit rehabilitation training group
Other: Strengthening, proprioceptive exercises. — -Strengthening exercise: Ankle Dorsiflexion and Plantar Flexion & inversion and eversion Strengthening with Exercise Bands
  -Proprioceptive exercise using wobble board
  Other Names: conventional physical therapy training

SUMMARY:
The goal of this clinical trial is to investigate the effect of Wii Fit rehabilitation on risk of fall, balance, and functional limitation, in patients with chronic ankle instability ,The main question it aims to answer is:

Are there any effect of Wii Fit rehabilitation training on balance, functional limitation, and risk of falls in patients with chronic ankle instability? Participants will be asked to sign a written informed consent form before the study according to guidelines of ethical committee The first group control group: 30 patients will receive conventional physical therapy training only which consist of strengthening, proprioceptive exercises.

The second group experimental group: 30 patients Wii Fit group will receive Wii Fit rehabilitation training and the same conventional exercise training.

DETAILED DESCRIPTION:
Wii Fit is an effective virtual reality approach for balance training. This intervention requires less time per session compared to traditional physical therapy treatment. Moreover, it is user-friendly, engaging, cost-effective and can be delivered at home without the need for supervision by a trained rehabilitation professional. Given the growing popularity of the technological approach as Wii Fit intervention, it would be important for the rehabilitation field to replicate these findings as high quality randomized clinical trials with large sample size and equal distribution of males and females.Further researches are needed to assess the long term effect of Wii training in patients with functional ankle instability. A variety of exercise programs were used as an intervention for chronic ankle instability, and conservative treatment interventions including balance, proprioceptive, and muscle strengthening exercises are effective for patients with chronic ankle instability

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients, their age ranges between 18 to 60 years old.
* Patients of both gender (men and women)
* A history of at least one ankle sprain, with the initial sprain occurring more than 1-year before the study
* A feeling of ''giving way'' at least 2 episodes in the last 6 months before the study
* Experiencing a recurring sprain, which is defined as two or more sprains on the same ankle
* No history of ankle injury within the three months prior to participation, and no cognitive deficit
* Capability to perform the intervention or daily activities without an increase in pain
* Currently they are not participating in any other rehabilitation exercise programs
* No history of ankle surgery

Exclusion Criteria:

* Subjects had balance deficits due to vestibular disorders, such as vertebro-basilar insufficiency and/or visual disorders
* Tumors in the area to be treated for the study
* pregnancy
* Any injury or surgery done in ankle joint, deformity at lower extremity
* Musculoskeletal condition like fracture, osteoporosis
* Neurological condition like parkinsonism disease, ataxia, stroke, muscular dystrophy, myasthenia gravis
* Cardiopulmonary conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Balance | "up to 8 weeks"
  will be assessed by Biodex balance system (overall, Anterior posterior and mediolateral balance indices with opened eyes and closed eyes).

SECONDARY OUTCOMES:
Functional limitation | "up to 8 weeks"
  will be assessed by Arabic version of the Foot and Ankle Ability Measure (FAAM). The FAAM consists of a 21-item Activities of Daily Living (ADL) scale and an 8- item Sports scale

OTHER OUTCOMES:
Risk of fall | "up to 8 weeks"
  will be assessed by the Arabic Version of the Falls Efficacy Scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: maher Ahmed el kablawy, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
NO individual participant data will be shared. Results will be published by the investigators in academic journal.
  sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators

REFERENCES:
- [Background] Punt IM, Armand S, Ziltener JL, Allet L. Effect of Wii Fit exercise therapy on gait parameters in ankle sprain patients: A randomized controlled trial. Gait Posture. 2017 Oct;58:52-58. doi: 10.1016/j.gaitpost.2017.06.284. Epub 2017 Jun 29. PMID 28735202
- [Background] Kim KJ, Heo M. Effects of virtual reality programs on balance in functional ankle instability. J Phys Ther Sci. 2015 Oct;27(10):3097-101. doi: 10.1589/jpts.27.3097. Epub 2015 Oct 30. PMID 26644652
- [Background] Kim KJ, Jun HJ, Heo M. Effects of Nintendo Wii Fit Plus training on ankle strength with functional ankle instability. J Phys Ther Sci. 2015 Nov;27(11):3381-5. doi: 10.1589/jpts.27.3381. Epub 2015 Nov 30. PMID 26696703
- [Background] Halaweh H, Svantesson U, Rosberg S, Willen C. Cross-Cultural Adaptation, Validity and Reliability of the Arabic Version of the Falls Efficacy Scale-International (FES-I). Med Princ Pract. 2016;25(1):1-7. doi: 10.1159/000441128. Epub 2015 Oct 20. PMID 26698595
- [Background] Franco JR, Jacobs K, Inzerillo C, Kluzik J. The effect of the Nintendo Wii Fit and exercise in improving balance and quality of life in community dwelling elders. Technol Health Care. 2012;20(2):95-115. doi: 10.3233/THC-2011-0661. PMID 22508022
- [Background] Afridi A, Malik AN, Ali S, Amjad I. Effect of balance training in older adults using Wii fit plus. J Pak Med Assoc. 2018 Mar;68(3):480-483. PMID 29540893
- [Background] Afridi A, Rathore FA, Nazir SNB. Wii Fit for Balance Training in Elderly: A Systematic Review. J Coll Physicians Surg Pak. 2021 May;31(5):559-566. doi: 10.29271/jcpsp.2021.05.559. PMID 34027869
- [Background] Alghadir AH, Iqbal ZA, Iqbal A, Ahmed H, Ramteke SU. Effect of Chronic Ankle Sprain on Pain, Range of Motion, Proprioception, and Balance among Athletes. Int J Environ Res Public Health. 2020 Jul 23;17(15):5318. doi: 10.3390/ijerph17155318. PMID 32718066
- [Background] Clark RA, Mentiplay BF, Pua YH, Bower KJ. Reliability and validity of the Wii Balance Board for assessment of standing balance: A systematic review. Gait Posture. 2018 Mar;61:40-54. doi: 10.1016/j.gaitpost.2017.12.022. Epub 2017 Dec 30. PMID 29304510
- [Background] Elsotohy NM, Salim YE, Nassif NS, Hanafy AF. Cross-education effect of balance training program in patients with chronic ankle instability: A randomized controlled trial. Injury. 2021 Mar;52(3):625-632. doi: 10.1016/j.injury.2020.09.065. Epub 2020 Oct 1. PMID 33041018
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1496-1505. doi: 10.1136/bjsports-2016-096189. Epub 2016 Jun 3. PMID 27259753
- [Background] Pourkazemi F, Hiller CE, Raymond J, Black D, Nightingale EJ, Refshauge KM. Predictors of recurrent sprains after an index lateral ankle sprain: a longitudinal study. Physiotherapy. 2018 Dec;104(4):430-437. doi: 10.1016/j.physio.2017.10.004. Epub 2017 Nov 2. PMID 29325691
- [Background] Seyedi M, Nobari H, Abbasi H, Khezri D, Oliveira R, Perez-Gomez J, Badicu G, Afonso J. Effect of Four Weeks of Home-Based Balance Training on the Performance in Individuals with Functional Ankle Instability: A Remote Online Study. Healthcare (Basel). 2021 Oct 23;9(11):1428. doi: 10.3390/healthcare9111428. PMID 34828475
- [Background] Shashidharan, Srisha & Selvan, Vijay. Effects of Virtual Reality Based Training (VRBT) and Proprioceptive Training for Improving Dynamic Balance in Chronic Ankle Instability (CAI) Patients -A Comparative Study (2022).
- [Derived] Abdel-Aal NM, El-Kablawy MA, Kadah MA, Abbas AAEH, Basha MA, Kamel FH. Effect of Wii Fit Rehabilitation on Balance, Functional Ability, and Risk of Falling in Patients With Chronic Ankle Instability: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2026 Feb 1;105(2):110-118. doi: 10.1097/PHM.0000000000002828. Epub 2025 Aug 13. PMID 40857124